CLINICAL TRIAL: NCT07056257
Title: The Effect of Adjunct Use of Diode Laser Therapy and Omega 3 Gel in Local Drug Delivery Approach on The Treatment of Localized Aggressive Periodontitis
Brief Title: Adjunct Use of Diode Laser Therapy and Omega 3 Gel in Local Drug Delivery Approach on The Treatment of Localized Aggressive Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dalia Mohammed Elsayed Ghannam, Dentist at ministry of health, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-OMPDR-4-22-11
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Diode Laser Therapy; Omega 3; Localized Aggressive Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Active Comparator): Thirteen sites [scaling-root planning (SRP)] were used as a control group.
  Interventions: Procedure: Scaling-root planning (SRP)
- Group II (Experimental): Thirteen sites [scaling-root planning (SRP)+ laser therapy with application of methyl cellulose gel at repeated times weekly for one month].
  Interventions: Procedure: Scaling-root planning (SRP)+ laser therapy
- Group III (Experimental): Thirteen sites [scaling-root planning (SRP) + omega 3 gel repeated time weekly for one month].
  Interventions: Procedure: Scaling-root planning (SRP)+ omega 3 gel
- Group IV (Experimental): Thirteen sites [combination therapy between scaling-root planning (SRP) + laser + omega 3 gel in repeated time weekly for one month].
  Interventions: Procedure: Scaling-root planning (SRP)+ laser therapy+ omega 3 gel

INTERVENTIONS:
Procedure: Scaling-root planning (SRP) — Thirteen sites [scaling-root planning (SRP)] were used as a control group.
  Arms: Group I
Procedure: Scaling-root planning (SRP)+ laser therapy — Thirteen sites [scaling-root planning (SRP)+ laser therapy with application of methyl cellulose gel at repeated times weekly for one month].
  Arms: Group II
Procedure: Scaling-root planning (SRP)+ omega 3 gel — Thirteen sites [scaling-root planning (SRP) + omega 3 gel repeated time weekly for one month].
  Arms: Group III
Procedure: Scaling-root planning (SRP)+ laser therapy+ omega 3 gel — Thirteen sites [combination therapy between scaling-root planning (SRP) + laser + omega 3 gel in repeated time weekly for one month].
  Arms: Group IV

SUMMARY:
This study aims to evaluate and compare the effect of combination therapy between diode laser and omega3 gel in the local drug delivery approach as an adjunct to scaling and root planning on the management of localized aggressive periodontitis clinically and immunologically.

DETAILED DESCRIPTION:
Periodontitis is a disease of the periodontium occurring in an otherwise healthy adolescent, which is characterized by a rapid loss of alveolar bone about more than one tooth of the permanent dentition.

The laser approach is an efficient and atraumatic technique to enhance its use for periodontal treatment. Within the limits of scientific data, treatment with diode laser and SRP showed a higher effect than SRP or laser alone.

Omega3 Polyunsaturated fatty acids (PUFA) have well recognized anti-inflammatory properties. They decrease inflammation through multiple pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with localized aggressive periodontitis.
* Patients must be medically free.
* Optimal compliance as evidenced by no missed treatment appointments and a positive attitude to maintain oral hygiene.
* Patients who are willing to participate in this study can enroll and complete it.

Exclusion Criteria:

* Patients with generalized aggressive periodontitis. Patients are over 35 years old.
* Pregnancy.
* Patients had scaling and root planning or antibiotic therapy in the last 6 months.
* Patients with hypersensitivity to fish oil.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Pocket depth | 6 months post-procedure
  Probing pocket depth (PD) was recorded according to Ramfijord 1967.

SECONDARY OUTCOMES:
Plaque score | 6 months post-procedure
  Plaque score was recorded according to Silness and loe 1964.
Bleeding on probing | 6 months post-procedure
  Bleeding on probing (BOP) according to Ainamo and Bay 1975.
Clinical attachment level loss | 6 months post-procedure
  Clinical attachment level loss (CAL) according to according to Ramfijord 1967.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.